CLINICAL TRIAL: NCT07298746
Title: OCT Angiography Changes of Retinal Microvasculature After Local Anesthesia in Cases Undergoing Cataract Surgery
Brief Title: Oct Angiography Changes After Local Anesthesia in Cataract Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amira Aldesoky Ahmed, Principal Investigator, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-25-9-22MS
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: OCTA Changes With Local Anesthesia
Keywords: OCTA , local anesthesia
MeSH Terms: interventions — Anesthesia, Local

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group A (Active Comparator): peribulbar anesthesia injection of two anesthetic agents ( lidocaine 2 %+ hyaluronidase 150IU\ML )
  Interventions: Drug: Local Anesthesia (peribular injection of both lidocaine 2 % and hyaluronidase 150IU\ML)
- group A1 (Active Comparator): peribulbar anesthesia injection ( mepivacaine 2% + hyaluronidase 150IU\ML )
  Interventions: Drug: Local Anesthesia (peribulbar anesthesia injection of mepivacaine 2% and hyaluronidase 150IU\ML)
- group B (Active Comparator): retrobulbar anesthesia injection ( lidocaine 2 %+ hyaluronidase 150IU\ML )
  Interventions: Drug: Local Anesthesia (retrobulbar anesthesia injection of lidocaine 2 % and hyaluronidase 150IU\ML)
- group B1 (Active Comparator): retrobulbar anesthesia injection ( mepivacaine 2% + hyaluronidase 150IU\ML )
  Interventions: Drug: local Anesthesia (retrobulbar anesthesia injection of mepivacaine 2% and hyaluronidase 150IU\ML)

INTERVENTIONS:
Drug: Local Anesthesia (peribular injection of both lidocaine 2 % and hyaluronidase 150IU\ML) — peribular injection of both lidocaine 2 % and hyaluronidase 150IU\ML
  Arms: group A
Drug: Local Anesthesia (peribulbar anesthesia injection of mepivacaine 2% and hyaluronidase 150IU\ML) — peribulbar anesthesia injection of mepivacaine 2% and hyaluronidase 150IU\ML
  Arms: group A1
Drug: Local Anesthesia (retrobulbar anesthesia injection of lidocaine 2 % and hyaluronidase 150IU\ML) — retrobulbar anesthesia injection of lidocaine 2 % and hyaluronidase 150IU\ML
  Arms: group B
Drug: local Anesthesia (retrobulbar anesthesia injection of mepivacaine 2% and hyaluronidase 150IU\ML) — retrobulbar anesthesia injection of mepivacaine 2% and hyaluronidase 150IU\ML
  Arms: group B1

SUMMARY:
Assessement of retinal microvasculature detected by OCT-angio after peribulbar &retrobulbar anesthesia in cases undergoing cataract surgery .

DETAILED DESCRIPTION:
prospective , interventional,comparative , clinical study utilizing a pre-post, within-subject design ,which will be conducted in the Department of Ophthalmology ,Sohag University Hospital ,Egypt.

Optical coherence tomography angiography (OCTA) will be performed before and after the administration of retrobulbar and peribulbar local anesthesia in the same cohort of patients, in order to evaluate the immediate effects of the anesthetic intervention on retinal microvascular parameters.the study will be conducted on patients aged 40-80 years with elective cataract surgery requiring regional block.the study will be divided into two main groups :

1. Group with peribulbar anesthesia injection.
2. Group with retrobulbar anesthesia injection.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged 40-80 years.
2. patients with elective cataract surgery requiring regional block.

Exclusion Criteria:

* 1.Allergy to study drugs. 2. Media opacities affecting OCT imaging (corneal pathologies, dense cataracts, vitreous.

opacities, etc). 3. Patients with any other retinal vascular diseases (retinal vein occlusion, central serous chorioretinopathy, age-related macular degeneration, etc).

4. Patients who have had previous intravitreal injections or Laser treatment. 5. Patients who underwent previous vitreoretinal surgeries. 6. Patients with uncontrolled glaucoma or ocular inflammations (eg: vitritis). 7.Patients with diabetes mellitus or hypertension.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Macular superficial capillary plexus (SCP) and deep capillary plexus (DCP | ntervention & data collection :4-6 monthes
  to detect degree of changes in vessel density at superficial and deep macular plexuses before and after injection of each group of anesthesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ali H, Eissa S, Magdy H, Khashba M. Dexmedetomidine as an Additive to Local Anesthesia for Decreasing Intraocular Pressure in Glaucoma Surgery: A Randomized Trial. Anesth Pain Med. 2020 Jun 27;10(3):e100673. doi: 10.5812/aapm.100673. eCollection 2020 Jun. PMID 32944557
- [Result] Rao HL, Pradhan ZS, Suh MH, Moghimi S, Mansouri K, Weinreb RN. Optical Coherence Tomography Angiography in Glaucoma. J Glaucoma. 2020 Apr;29(4):312-321. doi: 10.1097/IJG.0000000000001463. PMID 32053551
- [Result] Kalra G, Zarranz-Ventura J, Chahal R, Bernal-Morales C, Lupidi M, Chhablani J. Optical coherence tomography (OCT) angiolytics: a review of OCT angiography quantitative biomarkers. Surv Ophthalmol. 2022 Jul-Aug;67(4):1118-1134. doi: 10.1016/j.survophthal.2021.11.002. Epub 2021 Nov 5. PMID 34748794